CLINICAL TRIAL: NCT06946485
Title: A Clinical Study of the Safety and Efficacy of Universal Anti-CD70 CAR-T (CHT101) for the Treatment of Relapsed and Refractory Systemic Lupus Erythematosus
Brief Title: Universal Anti-CD70 CAR-T (CHT101) Cell Therapy for Relapsed Refractory Systemic Lupus Erythematosus
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHT101AIIT
Record Dates: First submitted 2025-04-02; First posted 2025-04-27 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-03

CONDITIONS: Systemic Lupus Erythematosus (SLE)
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Universal anti-CD70 CAR-T (CHT101) (Experimental)
  Interventions: Biological: Universal anti-CD70 CAR-T (CHT101)

INTERVENTIONS:
Biological: Universal anti-CD70 CAR-T (CHT101) — Universal anti-CD70 CAR-T (CHT101) cell therpy

SUMMARY:
This investigator-initiated trial aims to evaluate the safety and efficacy of universal anti-CD70 CAR-T (CHT101) in patients with relapsed refractory systemic lupus erythematosus.

DETAILED DESCRIPTION:
This study is a non-randomized, open-label, single-arm clinical trial designed to assess the efficacy and safety of universal anti-CD70 CAR-T (CHT101) in patients with relapsed refractory systemic lupus erythematosus.

ELIGIBILITY:
Inclusion Criteria:

1. Meet the 2019 EULAR/ACR classification criteria for systemic lupus erythematosus (SLE).
2. SLEDAI-2000 score >6.
3. Have at least one BILAG-2004 Grade A or two Grade B organ domain scores, or both.
4. Failure to respond to conventional therapy or disease relapse after remission. Conventional therapy: Glucocorticoids (≥1 mg/kg/day) combined with cyclophosphamide and ≥1 of the following immunosuppressants for >6 months: antimalarials, azathioprine, mycophenolate mofetil, methotrexate, leflunomide, tacrolimus, cyclosporine A, and/or biologics (e.g., rituximab, belimumab, telitacicept).
5. Aged 18-65 years; both genders eligible.
6. Adequate organ function:Bone marrow function: White blood cell count ≥3×10⁹/L. Absolute neutrophil count ≥1×10⁹/L (without colony-stimulating factor therapy within 2 weeks prior to testing). Hemoglobin ≥60 g/L; Liver function: Alanine aminotransferase (ALT) ≤3×upper limit of normal (ULN). Aspartate aminotransferase (AST) ≤3×ULN. Total bilirubin (TBIL) ≤1.5×ULN (except Gilbert's syndrome, TBIL ≤3.0×ULN); Renal function: Creatinine clearance (CrCl) ≥60 mL/min (calculated by Cockcroft-Gault formula); Coagulation: International normalized ratio (INR) ≤1.5×ULN. Prothrombin time (PT) ≤1.5×ULN; Cardiac function: Hemodynamic stability with left ventricular ejection fraction (LVEF) ≥55%.
7. Agrees to use double barrier methods, condoms, oral or injectable contraceptives, or intrauterine devices during the study period and for one year after taking the study medication. Females of childbearing potential must have a negative serum HCG test within 7 days prior to enrollment and must not be lactating.
8. Voluntarily participate in the study, provide written informed consent, and demonstrate good compliance with follow-up.

Exclusion Criteria:

1. Presence of neuropsychiatric lupus (NPSLE).
2. History of thrombotic thrombocytopenic purpura (TTP) or thrombotic microangiopathy (TMA).
3. History of severe drug allergies or hypersensitivity.
4. Active or suspected uncontrolled infections requiring treatment (including fungal, bacterial, viral, or other pathogens).
5. Central nervous system disorders caused by autoimmune diseases (ADs) or non-ADs.
6. Severe cardiac diseases.
7. Congenital immunoglobulin deficiency.
8. History of malignancy (except non-melanoma skin cancer, in situ cervical/bladder/breast/thyroid carcinoma with disease-free survival >5 years).
9. End-stage renal failure.
10. Participants meeting any of the following: Hepatitis B surface antigen (HBsAg)-positive or hepatitis B core antibody (HBcAb)-positive with detectable HBV DNA; Hepatitis C virus (HCV) antibody-positive with detectable HCV RNA; HIV antibody-positive; Syphilis-positive (RPR and TPHA positive, or TPHA positive with RPR reconfirmed positive after 4 weeks).
11. Psychiatric disorders or severe cognitive impairment.
12. Participation in other clinical trials within 3 months prior to enrollment.
13. Pregnant women or those planning pregnancy.
14. Other conditions deemed by the investigator to preclude study participation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
SRI-4 Response | SRI-4 response at 1 month after CHT101 infusion.
  SRI-4 Response defined as a decrease of ≥4 points from baseline in the SELENA-SLEDAI score, no new BILAG-evaluated grade A organs or <2 BILAG-evaluated grade B organs from baseline, and no deterioration in the physician's overall assessment (an increase of <0.30 points from baseline).
Safety Evaluation | safety evaluation Within 12 months after CHT101 infusion.
  Safety evaluation includes the collection of adverse events (AE), serious adverse events (SAE), vital signs and physical examinations, laboratory tests, including pregnancy tests and concomitant treatments. Safety is evaluated using the NCI-CTCAE 5.0 standard. CRS is evaluated using the ASTCT Consensus Grading Criteria, ICANS is evaluated using the Adult ASTCT ICANS Consensus Grading Criteria, acute GVHD is evaluated using the 2016 Mount Sinai Acute GVHD International Consortium Grading Criteria, and chronic GVHD is evaluated using the 2020 NCCN Hematopoietic Cell Transplantation Clinical Practice Guidelines, Version 1.0.

SECONDARY OUTCOMES:
Disease Activity Index | At 1 month, 2 month, 3 month, 6 month, 9 month, 12month after CHT101 infusion.
  The remission of SLE was based on the DORIS 2021 criteria, namely: SLEDAI=0 and PGA < 0.5 (0-3 points), serology was not considered, and patients could use antimalarial drugs, low-dose glucocorticoids (prednisolone ≤5mg/ day), and/or immunosuppressants including biologics.
Organ Damage | At 1 month, 2 month, 3 month, 6 month, 9 month, 12month after CHT101 infusion.
  The score was based on the SLE International Cooperation Group Injury Index (SDI). The higher the index, the worse the prognosis.
BILAG 2004 | At 1 month, 2 month, 3 month, 6 month, 9 month, 12month after CHT101 infusion.
  The absence of new organ Class A scores or two organ Class B scores indicates improvement.
Overall assessment of physicians | At 1 month, 2 month, 3 month, 6 month, 9 month, 12month after CHT101 infusion.
  The mitigation indicator was a baseline increase of less than 0.3 on a 3-point scale.

CONTACTS AND LOCATIONS:
Overall Officials: Lingyun Sun, Study Chair — The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Locations (1):
- The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School, Nanjing, Jiangsu, China